CLINICAL TRIAL: NCT01340300
Title: Randomized Phase II Study of Exercise and Metformin in Colorectal and Breast Cancer Survivors
Brief Title: Exercise and Metformin in Colorectal and Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey A. Meyerhardt, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-009
Record Dates: First submitted 2011-04-07; First posted 2011-04-22 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer; Breast Cancer
Keywords: Colorectal; Breast; Insulin; Exercise
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Insulin Resistance; Motor Activity | interventions — Exercise; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Exercise training (Active Comparator): Exercise training with exercise physiologist
  Interventions: Behavioral: Exercise training
- Exercise training with metformin (Active Comparator): Exercise training with exercise physiologist with oral metformin
  Interventions: Behavioral: Exercise training; Drug: Metformin
- Metformin (Active Comparator): Metformin
  Interventions: Drug: Metformin
- Control (Active Comparator): Educational information
  Interventions: Other: Educational information

INTERVENTIONS:
Behavioral: Exercise training — Two supervised exercise sessions per week
  Arms: Exercise training; Exercise training with metformin
Drug: Metformin — Oral metformin QD for two weeks, then BID
  Other Names: Fortamet, Glucophage, Glucophage XR, Glumetza, Riomet
  Arms: Exercise training with metformin; Metformin
Other: Educational information — educational information
  Arms: Control

SUMMARY:
Metformin is a medication that is commonly used in the treatment of diabetes. Recently small studies in cancer patients without diabetes suggest that metformin may benefit in lowering insulin levels. In those studies of patients with cancer but not diabetes, glucose (or sugar) levels in the blood are generally no lowered. Insulin and insulin-like growth factors affect the growth of cancer cells.

This randomized study will compare different interventions; exercise, exercise and metformin, metformin alone, or a control arm. The investigators are not directly testing how either exercise or metformin affects your disease. The investigators are testing how they affect insulin levels in your body as well as other blood markers. The investigators believe that these blood tests may either be related to cancer recurrences or be an early sign of cancer recurrences and they are testing how both exercise and metformin may change those markers.

DETAILED DESCRIPTION:
Subjects will be randomized into one of four groups: exercise training, exercise training and metformin, metformin alone, or control arm. All subjects will have lifestyle measurements, interviews regarding activity level, diet questionnaires, and blood tests.

Subjects randomized to exercise training will participate in two supervised exercise sessions per week with an exercise physiologist for 3 months. They will also be asked to exercise on their own for up to an additional 120 minutes each week.

Subjects randomized to exercise training and metformin will participate in two supervised exercise sessions per week and will take metformin. Metformin will be taken once daily for the first two weeks and then twice daily for 3 months.

Subjects randomized to metformin will take metformin once daily for the first two weeks and then twice daily.

Subjects on the control arm will receive a packet of educational information on nutrition and physical activity developed by the National Cancer Institute and American Cancer Society. In addition to education information, they will be offered two supervised sessions with an exercise physiologist as well as a pedometer 3 months after enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage I-III colorectal or breast cancer
* Undergone curative-intent complete surgical resection and completed all adjuvant therapy (if indicated) at least 2 months prior to enrollment
* Note: Breast cancer subjects on hormonal therapy or trastuzumab only therapy and colorectal cancer subjects on adjunctive therapies not considered cytotoxic chemotherapy (including those participating in CALGB 80702 receiving only celecoxib/placebo) are eligible.
* Participants will be allowed to receive concomitant adjuvant endocrine therapy for breast cancer; however, all endocrine agents must be initiated at least 1 month prior to enrollment in the study and continued throughout the duration of study participation.
* Less than 120 minutes of exercise per week
* Approval by oncologist or surgeon
* English speaking and able to read English
* No planned surgery anticipated in the 3 month intervention period
* At least one month from any major surgery to start of intervention including colostomy reversal

Exclusion Criteria:

* Concurrent other malignancy or history of other malignancy treated within the past 3 years (other than non-melanoma skin cancer or in-situ cervical cancer)
* Metastatic disease
* Scheduled to receive any form of further adjuvant cancer therapy
* Currently on medication for diabetes treatment
* Pregnant or breast-feeding
* Any condition associated with increased risk of metformin-associated lactic acidosis (prior renal failure or liver failure, history of acidosis of any type; habitual intake of 3 or more alcoholic beverages per day)
* Known hypersensitivity or intolerance to metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyerhardt, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Yale School of Medicine, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In a phase 2 RCT, stage I-III CRC & BC survivors at least 2 months from completing standard therapy were randomized. Major eligibility included absence of recurrence, absence of diabetes (glucose < 160 (random) or < 126 (fasting) mg/dl), and exercising < 120 min/wk. 1,426 patients screened, and 139 enrolled from September 2011 to December 2015.
Pre-assignment Details: Stratification factors: BMI (< 30 v > 30), gender, tumor site (CRC v BC)
Groups:
- Exercise Training With Metformin: Exercise training with exercise physiologist with oral metformin
  Exercise training plus metformin: Two supervised exercise sessions per week. Oral metformin QD for 2 weeks, then BID
Period: Overall Study
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
Started | 35 | 35 | 35 | 34
Baseline Blood Sample | 33 | 34 | 32 | 29
Follow-up Blood Sample | 25 | 26 | 19 | 18
Completed (Complete treatment and required follow-ups) | 26 | 26 | 20 | 20
Not Completed | 9 | 9 | 15 | 14
Not completed — Lost to Follow-up | 3 | 0 | 5 | 10
Not completed — Withdrawal by Subject | 5 | 6 | 6 | 3
Not completed — Adverse Event | 1 | 0 | 4 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Unrelated sickness | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control | Total
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 139
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [48 to 58] | 58 [49 to 65] | 55 [49 to 61] | 56 [48 to 66] | 55 [48 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 29 | 29 | 116
  Male | 6 | 6 | 6 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 31 | 35 | 34 | 33 | 133
  Unknown or Not Reported | 4 | 0 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 5 | 12
  White | 28 | 30 | 29 | 26 | 113
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 35 | 34 | 139
Study Site [Count of Participants; unit: Participants]
  DFCI | 28 | 22 | 24 | 25 | 99
  Duke | 4 | 4 | 5 | 6 | 19
  Yale | 3 | 9 | 6 | 3 | 21
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 27.7 [25.5 to 34.2] | 28.5 [26.4 to 32.8] | 28.8 [25.3 to 33.9] | 28.4 [25.5 to 31.9] | 28.5 [25.6 to 33.2]
Tumor Location [Count of Participants; unit: Participants]
  Breast Cancer | 22 | 21 | 22 | 22 | 87
  Colorectal Cancer | 13 | 14 | 13 | 12 | 52
Cancer Stage [Count of Participants; unit: Participants] — Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Participants
    stage I | 14 | 11 | 14 | 12 | 51
    stage II | 8 | 11 | 9 | 12 | 40
    stage III | 13 | 12 | 12 | 9 | 46
    Unknown stage | 0 | 1 | 0 | 1 | 2
Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 25 | 22 | 23 | 22 | 92
  No | 10 | 9 | 12 | 11 | 42
  Unknown | 0 | 4 | 0 | 1 | 5
Prior Radiation Therapy [Count of Participants; unit: Participants]
  Yes | 17 | 16 | 14 | 16 | 63
  No | 18 | 15 | 21 | 17 | 71
  Unknown | 0 | 4 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Insulin Level
Description: Determine whether supervised exercise training alone and metformin, either alone or in combination can decrease fasting insulin level from baseline to 3 months in patients who completed standard therapy for stage I-III colorectal or breast cancer. Fasting insulin levels in blood will be drawn at baseline, 3 months and 6 months. Negative least square means indicate a decrease at 3 month comparing to baseline value.
Time Frame: 0 and 3 months (change between 0 and 3 months)
Population: 11 patients are excluded for missing baseline blood samples.
Measure: Least Squares Mean (Standard Error); unit: mU/L
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
Number analyzed (Participants) | 33 | 34 | 32 | 29
mU/L | -2.47 (1.07) | -0.08 (1.06) | -1.16 (1.18) | 2.79 (1.27)
Statistical Analysis 1: Comparison: Exercise Training With Metformin vs Control; Null hypothesis: decrease of insulin in treatment arm is greater than the control arm; Test type: Superiority; p < 0.0001, Mixed Models Analysis — One-sided un-adjusted p-values to test if the decrease in treatment arm is greater than the control arm. Holm's method was performed for multiple comparisons to provide an overall significance level of 5%. Only significant p-values were reported; An intention-to-treat analysis, with a mixed model that was adjusted for baseline outcome value, BMI (< 30 or > 30), gender, cancer, and study site
Statistical Analysis 2: Comparison: Metformin vs Control; Null hypothesis: decrease of insulin in treatment arm is greater than the control arm; Test type: Superiority; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Exercise Training vs Control; Null hypothesis: decrease of insulin in treatment arm is greater than the control arm; Test type: Superiority; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Exercise Training With Metformin vs Metformin; Null hypothesis: decrease of Insulin in combined arm is greater than the exercise-only or metformin-only arm; Test type: Superiority; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Changes in Other Insulin-Related Biomarkers
Description: Markers related to insulin and insulin-like growth factors (including insulin-like growth factor 1 [IGF-1], IGF binding protein-1 [IGFBP-1], IGF binding protein-3 [IGFBP-3], leptin) will be measured by a blood draw at baseline, 3 months and 6 months. Negative least square means indicate a decrease at 3 month comparing to baseline value.
Time Frame: 0 and 3 months (change between 0 and 3 months)
Population: 11 patients are excluded for missing baseline blood samples.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
Number analyzed (Participants) | 33 | 34 | 32 | 29
ng/mL
  Leptin | -5.09 (1.21) | -0.54 (1.19) | -2.56 (1.33) | -0.20 (1.40)
  IGF-I | -1.29 (2.98) | 8.22 (2.94) | -2.66 (3.28) | -3.05 (3.46)
  IGFBP-1 | -0.22 (0.57) | 0.09 (0.56) | -1.20 (0.63) | 0.78 (0.66)
  IGFBP-3 | -178.8 (82.0) | 53.4 (80.7) | 25.9 (90.2) | -96.9 (94.9)
Statistical Analysis 1: Comparison: Exercise Training With Metformin vs Control; Null hypothesis: decrease of leptin in treatment arm is greater than the control arm; Test type: Superiority; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Metformin vs Control; Null hypothesis: decrease of IGFBP_1 in treatment arm is greater than the control arm; Test type: Superiority; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Exercise Training With Metformin vs Control; Null hypothesis: decrease of IGFBP_1 in treatment arm is greater than the control arm; Test type: Superiority; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Exercise Training With Metformin vs Exercise Training; Null hypothesis: decrease of Leptin in combined arm is greater than the exercise-only or metformin-only arm; Test type: Superiority; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Exercise Training With Metformin vs Metformin; Null hypothesis: decrease of Leptin in combined arm is greater than the exercise-only or metformin-only arm; Test type: Superiority; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Fasting Glucose Level
Description: Determine whether supervised exercise training alone and metformin, either alone or in combination can decrease fasting Glucose level from baseline to 3 months in patients who completed standard therapy for stage I-III colorectal or breast cancer. Fasting Glucose levels in blood will be drawn at baseline, 3 months and 6 months. Negative least square means indicate a decrease at 3 month comparing to baseline value.
Time Frame: 0 and 3 months (change between 0 and 3 months)
Population: 11 patients are excluded for missing baseline blood samples.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
Number analyzed (Participants) | 33 | 34 | 32 | 29
mg/dL | -0.09 (2.11) | 2.93 (2.08) | -4.11 (2.32) | 4.92 (2.44)
Statistical Analysis 1: Comparison: Metformin vs Control; Null hypothesis: decrease of Glucose in treatment arm is greater than the control arm; Test type: Superiority; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Exercise Training With Metformin vs Control; Null hypothesis: decrease of Glucose in treatment arm is greater than the control arm; Test type: Superiority; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Changes in Body Composition by Treatment Arm - Weight
Description: Negative least square means indicate a decrease at 3 month comparing to baseline value.
Time Frame: 0 and 3 months (change between 0 and 3 months)
Population: 2 patients are excluded for missing baseline measurements.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
Number analyzed (Participants) | 35 | 34 | 35 | 33
kg | -1.41 (0.53) | 0.70 (0.54) | -0.91 (0.57) | 1.97 (0.60)
Statistical Analysis 1: Comparison: Exercise Training With Metformin vs Control; Null hypothesis: decrease of Weight in treatment arm is greater than the control arm; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Metformin vs Control; Null hypothesis: decrease of Weight in treatment arm is greater than the control arm; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Exercise Training vs Control; Null hypothesis: decrease of Weight in treatment arm is greater than the control arm; Test type: Superiority; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

5. Other Pre Specified Outcome: Changes in Body Composition by Treatment Arm - BMI
Description: Negative least square means indicate a decrease at 3 month comparing to baseline value.
Time Frame: 0 and 3 months (change between 0 and 3 months)
Population: 2 patients are excluded for missing baseline measurements.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
Number analyzed (Participants) | 35 | 34 | 35 | 33
kg/m^2 | -0.51 (0.20) | 0.27 (0.20) | -0.33 (0.21) | 0.70 (0.22)
Statistical Analysis 1: Comparison: Exercise Training With Metformin vs Control; Null hypothesis: decrease of BMI in treatment arm is greater than the control arm; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Metformin vs Control; Null hypothesis: decrease of BMI in treatment arm is greater than the control arm; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Exercise Training vs Control; Null hypothesis: decrease of BMI in treatment arm is greater than the control arm; Test type: Superiority; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

6. Other Pre Specified Outcome: Changes in Body Composition by Treatment Arm - Waist to Hip Ratio
Description: Negative least square means indicate a decrease at 3 month comparing to baseline value.
Time Frame: 0 and 3 months (change between 0 and 3 months)
Population: 2 patients are excluded for missing baseline measurements.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
Number analyzed (Participants) | 35 | 34 | 35 | 33
ratio | -0.007 (0.01) | 0.006 (0.01) | 0.012 (0.01) | 0.016 (0.01)
Statistical Analysis 1: Comparison: Exercise Training With Metformin vs Control; Null hypothesis: decrease of Waist to Hip Ratio in treatment arm is greater than the control arm; Test type: Superiority; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Mortality was recorded for all patients. Non serious adverse events were collected for patients treated with Metformin (two arms: Exercise Training With Metformin, and Metformin only).
Arm/Group | Exercise Training With Metformin | Exercise Training | Metformin | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 21/35 | 0/0 | 23/35 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise Training With Metformin (N=35) | Exercise Training (N=0) | Metformin (N=35) | Control (N=0)
Diarrhea (Gastrointestinal disorders) | 8 | 0 | 12 | 0
Nausea (Gastrointestinal disorders) | 9 | 0 | 5 | 0
Abdomen Pain (Gastrointestinal disorders) | 6 | 0 | 6 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0 | 3 | 0
Bloating (Gastrointestinal disorders) | 3 | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 2 | 0
Headache (General disorders) | 1 | 0 | 1 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardiac disorders (Cardiac disorders) | 1 | 0 | 0 | 0
Dehydration (General disorders) | 0 | 0 | 1 | 0
Dry mouth (General disorders) | 0 | 0 | 1 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0
Hypertension (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypoglycemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypotension (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pain in extremity (General disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pharyngeal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Limited sample size, higher than anticipated dropout, short duration of therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes